CLINICAL TRIAL: NCT05094076
Title: Effect of Phosphate Exposure on Workers Respiratory and Oral Health in Phosphate Mine at Safaga
Brief Title: Effect of Phosphate Exposure on Workers Health
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mariam Roshdy Elkhayat, Principle investigator, Assiut University
Other Study IDs: Phosphate exposure
Record Dates: First submitted 2021-09-28; First posted 2021-10-26 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-09

CONDITIONS: Work-related Illness
MeSH Terms: interventions — X-Rays

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No

INTERVENTIONS:
Radiation: chest x ray — The chest radiographs obtained will be classiﬁed according to the International Labor Organization (ILO) System for Classiﬁcation of Radiographs for Pneumoconiosis [ILO, 1980]. Film quality, profusion, and shape and size of opacities will be evaluated by this method. Radiographic evidence of silicosis was deﬁned as a profusion score of 1/0 or greater
  Other Names: spirometer

SUMMARY:
To minimize negative health effects on health of workers in phosphate mining, it is important to assess, and diagnose health related effect of phosphate exposure & health hazards related to miners. Early reporting, diagnosis, and intervention can limit the severity of health hazards, improve the health services. To our knowledge no local previous studies were done in this area.

DETAILED DESCRIPTION:
Mining continues to be a dangerous activity, whether large-scale industrial mining or small-scale artisanal mining. Not only are there accidents, but exposure to dust and toxins, along with stress from the working environment or managerial pressures, give rise to a range of diseases that affect miners. Beneficiation is the process of removing the unnecessary minerals, which is used to increase the grade of mining product (concentrate). Phosphate ores can be beneficiated using one or a combination of different methods. The most common ones are: flotation, crushing, desliming, separation, grinding and washing thus keeping workers in Phosphate mines employ exposed to respirable dust pollution and to high silica dust levels presented in silicosis in many job areas, Silicosis is the most common occupational lung disease in Egypt where its prevalence rate ranges from 18.5 % to 45.8% among workers exposed to free crystalline silica dust. Despite its high prevalence, there is a lack of enforcement of exposure limits, availability and use of personal protective equipment, and occupational health education programs .

In Egyptian phosphate miners' study (2011), The study involved of three groups: 50 silica-exposed workers with radiological evidence of silicosis, 50 silica-exposed workers without evidence of silicosis, and 50 healthy unexposed subjects. , There were significant differences between pulmonary function parameters, values of C-reactive protein, rheumatoid factor, complement component C3, IgA, IgG, and IgM in exposed groups with and without silicosis, and healthy unexposed control subjects (p<.001).

Exposure to acid fumes in the phosphate mining was significantly associated with dental erosion and deteriorated oral health status, As working in phosphate mines had 8 and 28 times the risk for developing respectively oral lesions and teeth abrasions. This supported by Tunisian 2017 on 37 workers& 37 controls, found that frequencies of fluorosis, teeth abrasion, and oral lesions were significantly higher among the exposed group.

ELIGIBILITY:
Inclusion Criteria:

* Active working miners working in phosphate mines with minimum exposure 5 year.
* Had free pre-employment records.

Exclusion Criteria:

* Workers don't record phosphate exposure as in administration department.
* Workers with less than 5-year exposure
* Workers known to had autoimmune disorder before joining job.

Ages: 25 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Active working miners working in phosphate mines with minimum exposure 5 year.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2023-01-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
pneumoconiosis or not | through study completion, an average of 1 year
  The chest radiographs obtained will be classiﬁed according to the International Labor Organization (ILO) System for Classiﬁcation of Radiographs for Pneumoconiosis [ILO, 1980]. Film quality, profusion, and shape and size of opacities will be evaluated by this method. Radiographic evidence of silicosis was deﬁned as a profusion score of 1/0 or greater

SECONDARY OUTCOMES:
dental caries | through study completion, an average of 1 year
  The DMFT index is one of the simplest and most used indices in epidemiologic surveys of dental caries. It quantifies dental health status based on the number of carious, missing and filled teeth

REFERENCES:
- [Background] Stewart AG. Mining is bad for health: a voyage of discovery. Environ Geochem Health. 2020 Apr;42(4):1153-1165. doi: 10.1007/s10653-019-00367-7. Epub 2019 Jul 9. PMID 31289975
- [Background] Khelifi M, Zarrouk A, Nury T, Hamed H, Saguem S, Salah RB, Riedinger JM, Lizard G. Cytokine and eicosanoid profiles of phosphate mine workers. J Toxicol Sci. 2014 Jun;39(3):465-74. doi: 10.2131/jts.39.465. PMID 24849681
- [Background] Kalliny MS, Bassyouni MI. Immune response due to silica exposure in Egyptian phosphate mines. J Health Care Poor Underserved. 2011;22(4 Suppl):91-109. doi: 10.1353/hpu.2011.0156. PMID 22102308
- [Background] Amin WM, Al-Omoush SA, Hattab FN. Oral health status of workers exposed to acid fumes in phosphate and battery industries in Jordan. Int Dent J. 2001 Jun;51(3):169-74. doi: 10.1002/j.1875-595x.2001.tb00835.x. PMID 11563682